CLINICAL TRIAL: NCT01390766
Title: Drug Use Investigation for IMURAN (Azathioprine) Tablet (Hepatic Transplantation)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112305
Record Dates: First submitted 2011-06-23; First posted 2011-07-11 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Liver Diseases
Keywords: Antirejection
MeSH Terms: conditions — Liver Diseases | interventions — Azathioprine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed azathioprine tablet: Subjects prescribed azathioprine tablet during study period after the liver transplantation
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Azathioprine

SUMMARY:
This post-marketing surveillance (PMS) study is designed to investigate the efficacy and safety of azathioprine tablets in Japanese subjects whom liver transplantation is performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who undergo liver transplantation and azathioprine tablet was administered

Exclusion Criteria:

As this is PMS study, there are no exclusion criteria but contraindications are as follows.

* Subjects with hypersensitivity to the ingredients of azathioprine tablet
* Subjects who is pregnant or might be pregnant
* Subjects whose white count is lower than 3000/cubic millimeter

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The following subjects to whom azathioprine tablet is administered for "the suppression of liver transplant rejection";
  * Subjects on whom liver transplantation is performed and to whom azathioprine tablet is administered within 1 year after transplant surgery from the approval date of the additional indication of azathioprine tablet for liver transplantation (20 June 2001) to May 2010.
  * Subjects on whom liver transplantation is performed before the approval date of the additional indication of azathioprine tablet for liver transplantation (20 June 2001) and to whom azathioprine tablet is administered within 1 year after transplant surgery.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2002-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events related to azathioprine tablets and serious adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline